CLINICAL TRIAL: NCT04469907
Title: A Single Dose, Non-Randomized, Open-Label, Parallel Group Study to Assess the Pharmacokinetics, Safety and Tolerability of AZD9977 in Participants With Renal Impairment
Brief Title: Study to Assess the Pharmacokinetics and Safety of AZD9977 in Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6401C00008
Record Dates: First submitted 2020-06-19; First posted 2020-07-14 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — AZD9977

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment - AZD9977 (Experimental): There are 4 cohorts in this arm based on renal function (mild, moderate, severe, and normal). Each cohort will have 8 participants.
  Interventions: Drug: AZD9977

INTERVENTIONS:
Drug: AZD9977 — Participants will receive a single oral dose of AZD9977 under fasted conditions.

SUMMARY:
This is a single dose, non-randomized, open-label, parallel group study. The study will be conducted in participants with severe renal impairment and compared with matched participants with normal renal function. The duration of the study for an individual participant from Screening to Follow-up will be approximately 5 weeks.

DETAILED DESCRIPTION:
The study will have 4 cohorts, consisting of participants with severe renal impairment who are not on dialysis (Cohort 1), moderate renal impairment (Cohort 2), mild renal impairment (Cohort 3) and participants with normal renal function (Cohort 4). Following completion of Cohort 1 and Cohort 4, pharmacokinetics (PK) and safety data will be reviewed and a decision will be made whether to study unmatched participants with moderate and mild renal impairment (Cohorts 2 and 3, respectively).

Participants will be screened up to 21 days before administration of study drug. Eligible participants will be admitted to the clinical unit either on the evening of Day -2 or on the morning of Day -1. Each participant will receive a single oral dose of the study drug under fasted conditions on Day 1. Participants will be required to remain resident in the clinical unit until the morning of Day 3 but, if participants prefer, may also remain resident until all PK and other study procedures are completed on Day 7. This decision to extend residency will be made at the discretion of the principal investigator. If participants do check out on Day 3, participants will then return to the unit, as scheduled, for collection of PK samples and safety assessments, with a final Follow-up Visit on Day 14.

ELIGIBILITY:
Inclusion Criteria:

Healthy matched control participants only (Cohort 4):

1. Participants who are overtly healthy.
2. Stable renal function, with eGFR of ≥ 90 mL/min/1.73m^2.

   Renally impaired participants only (Cohorts 1-3):
3. Participants who have renal impairment:

   1. Cohort 1 participants with severe renal impairment must have an eGFR lesser than 30 mL/min/1.73m^2 not on dialysis
   2. Cohort 2 participants with moderate renal impairment must have an eGFR of greater than or equal to 30 to lesser than 60 mL/min/1.73m^2
   3. Cohort 3 participants with mild renal impairment must have an eGFR of greater than or equal to 60 to lesser than 90 mL/min/1.73m^2.

   All participants (Cohorts 1-4):
4. Body weight of at least 50 kg and BMI within the range greater than or equal to 18 to lesser than or equal to 35 kg/m^2.
5. Male or female of non-childbearing potential.
6. Male participants should not donate sperm for the duration of the study.
7. Female participants must have a negative pregnancy test at time of study entry.
8. Capable of giving signed informed consent.

Exclusion Criteria:

Healthy matched control participants only (Cohort 4):

1. Evidence of clinically significant cardiovascular, hematological, renal, endocrine, pulmonary, gastrointestinal, hepatic, neurologic, psychiatric, inflammatory or allergic disease.

   Renally impaired participants only (Cohorts 1-3):
2. Renal transplant participants, participants on dialysis and those with a history of acute kidney injury.

   All participants (Cohorts 1-4):
3. Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus antibody.
4. Known history of drug or alcohol abuse.
5. History of QT prolongation and arrhythmia.
6. Any moderate or potent inhibitors or inducers of CYP3A4.
7. Participants with a known hypersensitivity to AZD9977 or any of the excipients of the product.
8. For women only - currently pregnant or breast-feeding.
9. A positive local diagnostic test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening, clinical signs and symptoms consistent with COVID-19, or the patient has been previosuly hospitalised with COVID-19 infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Area under the plasma concentration-time curve from time zero to infinity (AUC) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC0-t) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Time to reach maximum observed plasma concentration (tmax) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Half-life associated with terminal slope of a semi-logarithmic concentration time curve (t½λz) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Terminal elimination rate constant (λz) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Apparent total body clearance of drug from plasma after oral administration (CL/F) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Non-renal clearance of drug from plasma after oral administration (CLNR/F) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Apparent volume of distribution during the terminal phase after oral administration (Vz/F) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Mean residence time (MRT) | Day 1 to 3 (Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 20, 24, 36, and 48 hours post-dose), Day 4 to 7
  To assess the PK of AZD9977 following administration of AZD9977
Renal clearance of the drug from plasma (CLR) | Day 1 to 3 (Pre-dose, 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-dose)
  To assess the PK of AZD9977 following administration of AZD9977
Cumulative amount of unchanged drug excreted into the urine (Ae) | Day 1 to 3 (Pre-dose, 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-dose)
  To assess the PK of AZD9977 following administration of AZD9977
Fraction of the drug excreted into the urine (fe) | Day 1 to 3 (Pre-dose, 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-dose)
  To assess the PK of AZD9977 following administration of AZD9977

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Day -2 to Day 14
  To evaluate the safety and tolerability of AZD9977
Estimated Glomerular Filtration Rate (eGFR) | Screening, Day -1, Day 1 to 3 (Pre-dose, 4, 12, 24 , 36, and 48 hours)
  To determine eGFR based on creatinine and cystatin C using CKD-EPI formula

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, Northridge, California
  - Research Site, DeLand, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Blue Ash, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home